CLINICAL TRIAL: NCT01907789
Title: Prophylactic Salpingectomy With Delayed Oophorectomy, Risk-Reducing Salpingo-Oophorectomy, and Ovarian Cancer Screening Among BRCA Mutation Carriers: A Proof-of-Concept Study
Brief Title: Prophylactic Salpingectomy With Delayed Oophorectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-0340; NCI-2015-00465 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-18; First posted 2013-07-25 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian Carcinoma; Ovary; BRCA Mutation Carriers; BRCA1 or BRCA2 mutation; High risk for developing ovarian cancer; Ovarian cancer screening; Risk-reducing salpingo-oophorectomy; RRSO; Prophylactic salpingectomy with delayed oophorectomy; PSDO; Questionnaire; Quality of life; QOL; Survey; Transvaginal ultrasound; Phone call
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ovarian Cancer Screening (Experimental): Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer will return to clinic every six months to undergo screening for ovarian cancer symptoms, physical examination, CA125, HE4, and transvaginal ultrasound.
  Interventions: Other: Ovarian Cancer Screening; Behavioral: Questionnaire; Procedure: Transvaginal Ultrasound; Behavioral: Phone Call
- Prophylactic Salpingectomy with Delayed Oophorectomy (PSDO) (Experimental): Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer have salpingectomy performed as an outpatient procedure. After the 3-year follow up period, oophorectomy performed as an outpatient procedure.
  Interventions: Procedure: Prophylactic Salpingectomy with Delayed Oophorectomy; Behavioral: Questionnaire; Procedure: Transvaginal Ultrasound; Behavioral: Phone Call
- Risk-Reducing Salpingo-Oophorectomy (RRSO) (Experimental): Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer have risk-reducing salpingo-oophorectomy (RRSO) performed as an outpatient procedure.
  Interventions: Procedure: Risk-Reducing Salpingo-Oophorectomy; Behavioral: Questionnaire; Procedure: Transvaginal Ultrasound; Behavioral: Phone Call

INTERVENTIONS:
Other: Ovarian Cancer Screening — Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer will return to clinic every six months to undergo screening for ovarian cancer symptoms, physical examination, CA125, HE4, and transvaginal ultrasound.
  Arms: Ovarian Cancer Screening
Procedure: Prophylactic Salpingectomy with Delayed Oophorectomy — Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer have salpingectomy performed as an outpatient procedure. After the 3-year follow up period, oophorectomy performed as an outpatient procedure.
  Arms: Prophylactic Salpingectomy with Delayed Oophorectomy (PSDO)
Procedure: Risk-Reducing Salpingo-Oophorectomy — Woman who have a mutation (genetic change) in one of the BRCA genes, and are at high risk for developing ovarian cancer have risk-reducing salpingo-oophorectomy (RRSO) performed as an outpatient procedure.
  Arms: Risk-Reducing Salpingo-Oophorectomy (RRSO)
Behavioral: Questionnaire — Ovarian Screening Group: Quality of life (QOL) questionnaire completed at baseline, end of year 1, 2, and 3.
  Prophylactic Salpingectomy with Delayed Oophorectomy (PSDO): Quality of life (QOL) questionnaire completed at baseline, 1 month 1 year, 2 years, and 3 years after salpingectomy. Also before oophorectomy performed, 1 month and 6 months after oophorectomy.
  Risk-Reducing Salpingo-Oophorectomy (RRSO) Group: Quality of life (QOL) questionnaire completed at baseline, then 1 month, 6 months, and 1 year after surgery.
  Other Names: Survey
Procedure: Transvaginal Ultrasound — Ovarian Cancer Screening Group: Transvaginal ultrasound performed at baseline and every 6 months for 3 years.
  Prophylactic Salpingectomy with Delayed Oophorectomy (PSDO) group: Transvaginal ultrasound performed at baseline, every 6 months for 3 years after salpingectomy, then before oophorectomy.
  Risk-Reducing Salpingo-Oophorectomy (RRSO) Group: Transvaginal ultrasound performed at baseline.
Behavioral: Phone Call — Ovarian Cancer Screening Group and Prophylactic Salpingectomy with Delayed Oophorectomy (PSDO) Group: Phone call made to patient one time a year after third year follow up.
  Risk-Reducing Salpingo-Oophorectomy (RRSO) Group: Phone call made to patient 1 day after surgery, 1 week after surgery, then yearly.

SUMMARY:
The goal of this clinical research study is to compare ovarian cancer screening, risk-reducing salpingo-oophorectomy (RRSO), and prophylactic salpingectomy with delayed oophorectomy (PSDO). The safety of RRSO and PSDO will also be studied.

Ovarian cancer screening does not involve a surgical procedure. Instead, physical exams, blood tests, and ultrasound are used to check for ovarian, fallopian tube, and peritoneal cancer.

The surgical procedures, RRSO and PSDO, are designed to lower your risk of ovarian cancer.

In RRSO, the fallopian tubes and ovaries are removed at the same time.

In PSDO, the fallopian tubes are removed and the ovaries remain in place so that the patient does not go through menopause. The ovaries are removed at a later date. The main goal of this study is to learn how many patients actually have their ovaries removed at a later date. Researchers also want to learn whether the removal of fallopian tubes will decrease the risk of ovarian cancer.

DETAILED DESCRIPTION:
This study has 3 options: ovarian cancer screening, PSDO, and RRSO. You may choose which study group you want to take part in. However, you must let the researchers know what your choice is before any testing for the study begins. The 3 study groups are described in detail below.

GROUP 1: OVARIAN CANCER SCREENING:

Study Visits:

For this group, there is no testing required before starting the study. If you agree to be in Group 1, the following tests and procedures will be performed:

* You will have a physical exam, including a pelvic exam.
* You will have a transvaginal ultrasound (ultrasound inside the vagina) to look at your ovaries and fallopian tubes.
* Blood (about 2 tablespoons) will be drawn to measure your CA125 levels. This test is used to screen for ovarian cancer.
* You will complete a questionnaire about your quality of life. This should take up to 15 minutes.

Every 6 months for up to 3 years:

* You will have a physical exam, including a pelvic exam.
* Blood (about 2 tablespoons) will be drawn for CA-125 testing.
* You will have a transvaginal ultrasound to look at your ovaries and fallopian tubes.

At the end of Years 1, 2, and 3, you will complete the quality-of-life questionnaire.

All of your test results will be discussed with you. If any of your test results are abnormal, the study doctor may ask you to have additional testing, which may include CA-125 testing, ultrasound, and/or a computed tomography (CT) scan or magnetic resonance imaging (MRI). If the results show cancer, the study doctor will refer you to a gynecologic oncologist (a doctor for women's cancer) and/or recommend that you have your ovaries and fallopian tubes removed.

Length of Study:

You may have study visits for up to 3 years. You will be taken off study early if you develop cancer or if you are unable to follow study directions.

At any time or preferably at the end of 3 years, you will have the option to cross over and choose one of the treatment options (Group 2 or 3).

Follow-Up:

One (1) time a year after your last study visit for as long as needed, the study staff will contact you by phone, e-mail, or letter to ask if you have had any changes in your medical history. If you are called, the calls should last about 5 minutes.

GROUP 2: FALLOPIAN TUBE REMOVAL WITH DELAYED OVARY REMOVAL (PSDO):

Salpingectomy:

If you are found to be eligible to take part in this study in Group 2, the study doctor will discuss the salpingectomy surgery with you in detail, including the risks and possible benefits. You will be asked to sign a surgical consent form. After that, the salpingectomy will be scheduled.

Most patients have salpingectomy performed as an outpatient procedure. This means that you will likely go home the day of your surgery. If the study doctor plans to have you stay overnight in the hospital for any reason, it will be discussed with you.

During the surgery, the inside of your abdomen will be looked at and both of your fallopian tubes will be removed. If the study doctor finds anything during the surgery that may be cancerous, a tissue sample or a complete ovary will be removed during surgery and tested. If cancer is found, a gynecologic oncologist would perform your cancer surgery.

Post-Salpingectomy Follow-Up:

The study staff will call you 1 day and 1 week after surgery to ask how you are doing. The calls should last about 5 minutes.

One (1) month after surgery:

* You will have a physical exam, including an exam of your surgical incisions (wounds).
* You will complete the quality-of-life questionnaire.

The pathology (tissue) results from your surgery will be discussed with you at either the 1-week phone call or the 1-month visit. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

Ovarian Cancer Screening Period:

Every 6 months or until your delayed oophorectomy after the salpingectomy:

* You will have a physical exam, including a pelvic exam.
* Blood (about 2 tablespoons) will be drawn for CA-125 testing.
* You will have a transvaginal ultrasound to look at your ovaries.

You will complete the quality-of-life questionnaire 1 time a year until 1 year after your delayed oophorectomy.

Pre-Oophorectomy Testing:

After the 3-year screening period, you will have a pre-oophorectomy visit. The following tests and procedures will be performed:

* You will have a physical exam, including a pelvic exam.
* Blood (about 2 tablespoons) will be drawn for routine tests and CA-125 testing.
* You will have a transvaginal ultrasound to look at your ovaries, if this has not been done in the last 6 months.
* You will complete the quality-of-life questionnaire, if this has not been done in the last 6 months.
* You may have other tests performed if the study doctor thinks it is needed.

Oophorectomy:

If your pre-surgical testing is normal, the study doctor will discuss the planned surgery with you in detail, including the risks and possible benefits. You will be asked to sign a surgical consent form. After that, the oophorectomy will be scheduled.

Most patients have oophorectomy performed as an outpatient procedure. This means that you will likely go home the day of your surgery. If the study doctor plans to have you stay overnight in the hospital for any reason, it will be discussed with you.

During the surgery, the inside of your abdomen will be looked at and both of your ovaries will be removed. If the study doctor finds anything during the surgery that may be cancerous, a tissue sample will be removed during surgery and tested.

Post-Oophorectomy Follow-Up:

The study staff will call you 1 day and 1 week after surgery to ask how you are doing.

One (1) month after surgery:

* You will have a physical exam, including an exam of your surgical incisions.
* You will complete the quality-of-life questionnaire.

The pathology results from your surgery will be discussed with you at either the 1-week phone call or the 1-month visit. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

At 6 months and 1 year after surgery, you will complete the quality-of-life questionnaire.

At 1 year after surgery:

* You will have a physical exam, including a pelvic exam.
* Blood (about 2 tablespoons) will be drawn for CA-125 testing.

All of your test results will be discussed with you. If any of your test results are abnormal, the study doctor may ask you to have additional testing, which may include CA-125 testing, ultrasound, and/or a CT scan or MRI. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

Length of Study:

You will have study visits until 1 year after your oophorectomy. You will be taken off study early if you develop cancer or if you are unable to follow study directions.

Follow-Up:

One (1) time a year after your last study visit for as long as needed, the study staff will contact you by phone, e-mail, or letter to ask if you have had any changes in your medical history.

GROUP 3: REMOVAL OF FALLOPIAN TUBES AND OVARIES AT THE SAME TIME (RRSO):

RRSO:

If you are found to be eligible to take part in this study in Group 3, the study doctor will discuss the surgery with you in detail, including the risks and possible benefits. You will be asked to sign a surgical consent form. After that, the RRSO will be scheduled.

Most patients have RRSO performed as an outpatient procedure. This means that you will likely go home the day of your surgery. If the study doctor plans to have you stay overnight in the hospital for any reason, it will be discussed with you.

During the surgery, the inside of your abdomen will be looked at and both of your ovaries and fallopian tubes will be removed. If the study doctor finds anything during the surgery that may be cancerous, a tissue sample will be removed during surgery and tested.

The pathology results from your surgery will be discussed with you at either the 1-week phone call or the 1-month visit. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

Post-Surgery Follow-Up:

The study staff will call you 1 day and 1 week after surgery to ask how you are doing.

One (1) month after surgery:

* You will have a physical exam, including an exam of your surgical incisions.
* You will complete the quality-of-life questionnaire.

The pathology results from your surgery will be discussed with you at either the 1-week phone call or the 1-month visit. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

At 6 months and 1 year after surgery, you will complete the quality-of-life questionnaire.

At 1 year after surgery:

* You will have a physical exam, including a pelvic exam.
* Blood (about 2 tablespoons) will be drawn to measure your CA-125.

All of your test results will be discussed with you. If any of your test results are abnormal, the study doctor may ask you to have additional testing, which may include CA-125 testing, ultrasound, and/or a CT scan or MRI. If the results show cancer, the study doctor will refer you to a gynecologic oncologist.

Length of Study:

You will have study visits for up to 1 year after surgery. You will be taken off study early if you develop cancer or if you are unable to follow study directions.

Follow-Up:

One (1) time a year after your last study visit for as long as needed, the study staff will contact you by phone, e-mail, or letter to ask if you have had any changes in your medical history.

This is an investigational study. At this time, the only known method that may lower your risk of ovarian cancer is to have both of your ovaries and fallopian tubes removed (RRSO). Screening for ovarian cancer does not lower the risk that you will develop cancer. PSDO has not previously been studied and may not lower your ovarian cancer risk. PSDO is currently being used for research purposes only.

Up to 80 women will take part in this multicenter study. Up to 60 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women with a documented BRCA1 or BRCA2 mutation. Menopause is defined as >/= 12 months of amenorrhea.
2. Women must be at least 30 and less than 48 years of age.
3. Candidate for surgery and willing to undergo two surgical procedures (if chooses the PSDO arm).
4. Patient choosing PSDO or RRSO must desire permanent sterilization.
5. Presence of at least one fallopian tube. Prior tubal ligation is allowed.
6. Participants may have a personal history of non-ovarian malignancy, but must be without evidence of disease at enrollment and the patient must have completed treatment (including surgery, chemotherapy, or radiotherapy) > 3 months prior to enrollment (other than non-melanoma skin cancer). Current or past SERM or aromatase inhibitor use is allowed.
7. Willingness to return to the enrolling site for any surgical procedures including pre-operative and post-operative care.
8. Willingness to return to the enrolling site for ovarian cancer screening during the study period.

Exclusion Criteria:

1. Postmenopausal women or women < 30 or >/= 48 years of age.
2. Women without a documented BRCA mutation.
3. Women with a history of ovarian, fallopian tube, or primary peritoneal cancer.
4. Women currently undergoing cancer treatment or with a known active cancer. History of malignancy is allowed as long as the patient has completed treatment > 3 months prior to enrollment.
5. Medical comorbidities making surgery unsafe as determined by the patient's surgeon.
6. Prior bilateral salpingectomy. Prior unilateral salpingectomy is allowed.
7. Women who are pregnant. Patients are deemed not pregnant by virtue of urine pregnancy test (UPT), transvaginal ultrasound, beta HCG, or best judgement of the investigator. Pregnancy testing is not required per protocol to determine study eligibility.
8. Women desiring future fertility except in the screening arm of the trial.
9. Women whose most recent CA125 or transvaginal ultrasound is abnormal. A history of abnormal CA125 or ultrasound is allowed, as long as the most recent testing is normal.
10. Inability to provide informed consent.
11. Inability to read or speak English.

Ages: 30 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-08-26 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Compliance with Prophylactic Salpingectomy with Delayed Oophorectomy Strategy | Up to 5 years
  The proportion of women who comply with the prophylactic salpingectomy with delayed oophorectomy strategy estimated with an exact 95% binomial confidence interval. If all 20 patients return for their scheduled oophorectomy the 95% confidence interval for the proportion of women who are compliant will be 0.846 to 1.00.

SECONDARY OUTCOMES:
Number of occult malignancies | Up to 5 years
  Will be tabulated by study arm. The risk difference will be estimated for occult malignancies with 95% confidence intervals, where the risk is defined as the number of events divided by the total time at risk.
Number of complications | Up to 5 years
  Will be tabulated by study arm. The risk difference will be estimated for complications with 95% confidence intervals, where the risk is defined as the number of events divided by the total time at risk.
Type of complications | Up to 5 years
  Will be tabulated by study arm. The risk difference will be estimated for complications with 95% confidence intervals, where the risk is defined as the number of events divided by the total time at risk.
Change in quality of life measure | Baseline to up to 3 years
  Descriptive statistics and box plots will be used to summarize the quality of life measures at each assessment time for each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Nebgen, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - NorthShore University Health System, Evanston, Illinois
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org